CLINICAL TRIAL: NCT00299676
Title: An Observational Study of Clinical Outcomes and Safety Profile of Galantamine in the Treatment of Patients With Alzheimer's Disease Over an 18-month Period
Brief Title: An Observational Study of the Safety and Effectiveness of Galantamine in the Treatment of Patients With Alzheimer's Disease Over an 18-month Period
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CR004816
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Alzheimer Disease; Dementia; Galantamine
Keywords: Alzheimer's Disease; Dementia; Post Marketing; Prospective Studies; Longitudinal Studies; New Zealand; Cholinesterase Inhibitors; Observational; Outcomes
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Galantamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001: Galantamine (Reminyl) Use of Reminyl according to approved NZ data sheet
  Interventions: Drug: Galantamine (Reminyl)

INTERVENTIONS:
Drug: Galantamine (Reminyl) — Use of Reminyl according to approved NZ data sheet

SUMMARY:
The purpose of this observational study is to investigate the changes in cognitive functioning, behavior, and functional improvement in Alzheimer's disease patients treated with Galantamine who are living at home (i.e. not in permanent residential care), and to obtain information regarding usual clinical practice that can be used for communicating treatment expectations to patients and supporters.

DETAILED DESCRIPTION:
This is a prospective, observational study to assess the changes in cognitive functioning, behavior, and functional improvement in Alzheimer's disease patients treated with Galantamine who are living at home (i.e. not in permanent residential care), and to obtain information regarding usual clinical practice performed by relevant specialists. There will be no experimental component associated with this study and all observational activities will be part of routine care. This study will follow patients with Alzheimer's disease, who are currently not in permanent residential care, for a period of 18 months. The three domains of cognition, behavior and function will be evaluated at baseline using the Mini-Mental State Examination (MMSE) and/or ADAS-Cog, the abridged Instrumental Activities of Daily Living (IADL) and a 14-item behavioral assessment scale. Changes in the 3 domains will be observed after 3, 6, 12 and 18 months of Galantamine therapy through the completion of The Clinician Interview Based Impression of Change (CIBIC-Plus), abridged IADL, behavioral changes, and the Mini-Mental State Examination/ADAS-Cog. Primary outcome is to determine changes from baseline in cognition, behavior and function will be assessed after 3, 6, 12, and 18 months as measured by the CIBIC-Plus, abridged IADL, the Mini-Mental State Examination/ADAS-Cog and behavioral changes. The secondary outcome is development of information regarding treatment expectations that can be used for communicating with patients and supporters. Galantamine will be prescribed according to routine clinical practice and as per the Product Information leaflet

ELIGIBILITY:
Inclusion Criteria:

* Patients prescribed with galantamine according to the approved New Zealand Data Sheet
* The clinical decision to prescribe Galantamine must have been made before and independently of the decision to enroll the patient in this observational study
* The patient should not have commenced Galantamine treatment before the baseline visit
* Patients must be currently living at home (i.e. not in permanent residential care)
* Availability of a supporter who has regular contact with the patient

Exclusion Criteria:

* Patients having known hypersensitivity to Galantamine
* Having severe liver impairment or severe kidney impairment
* Suffering from an uncontrolled medical condition other than dementia
* Being treated, or previously treated, with another cholinesterase inhibitor or other cholinomimetics (medications for treating Alzheimer's disease)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Alzheimer's disease, who are currently not in permanent residential care. A convenience sampling method was applied.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2005-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Investigate the change in cognitive functioning, clinical and functional improvement, in patients treated with REMINYL in a naturalistic setting. | Baseline, month 3, month 6, month 12 and month 18.

SECONDARY OUTCOMES:
Development of information regarding treatment expectations that can be used for communicating with patients and supporters. | Baseline, month 3, month 6, month 12 and month 18.
Gain usage experience in a clinical practice setting that can be used for communicating treatment expectations to patients and carers. | Baseline, month 3, month 6, month 12 and month 18.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pty Ltd Clinical Trial, Study Director — Janssen-Cilag Pty Ltd
Locations (5):
- Australia (5):
  - Auckland
  - Christchurch Nz
  - Hamilton
  - Porirua
  - Tauranga